CLINICAL TRIAL: NCT04284254
Title: Sleeping Beauty Transposon-Engineered Plasmablasts for Expression and Delivery of Alpha-L-iduronidase in Patients With Hurler Syndrome That Have Previously Undergone Allogeneic Transplantation
Brief Title: MT2018-18: Sleeping Beauty Transposon-Engineered Plasmablasts for Hurler Syndrome Post Allo HSCT
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study went on hold because more pre-clinical work needs to be done per FDA feedback. However, the study never went off hold and the study team has decided to close this study without opening to enrollment.
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2018LS094; MT2018-18 (Other: University of Minnesota Masonic Cancer Center)
Record Dates: First submitted 2019-11-11; First posted 2020-02-25 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: Mucopolysaccharidosis Type IH (MPS IH, Hurler Syndrome); Mucopolysaccharidosis Type IH; MPS IH, Hurler Syndrome
Keywords: MPS IH; Hurler syndrome
MeSH Terms: conditions — Mucopolysaccharidosis I | interventions — sleeping beauty transposase, human

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Phase 1: Dose Escalation (Experimental)
  Interventions: Drug: Autologous Plasmablasts
- Phase 2 - Expansion at MTD (Experimental)
  Interventions: Drug: Autologous Plasmablasts

INTERVENTIONS:
Drug: Autologous Plasmablasts — Autologous Plasmablasts engineered to express α-L-iduronidase (IDUA) using the Sleeping Beauty transposon system.
  Phase 1:
  * Dose Level 1: 5 x 10e7 cells/kg on Day 0
  * Dose Level 2: 1 x 10e8 cells/kg on Day 0
  * Dose Level 3: 1 x 10e8 cells/kg x 2 doses on Day 0 and Day 30 +/-3 days.
  Phase 2:
  - Maximum Tolerated Dose (MTD) established in Phase I
  Other Names: Sleeping Beauty

SUMMARY:
This is a single center, Phase 1/2 study in which patients with Hurler syndrome who have previously undergone allogeneic hematopoietic stem cell transplantation are treated with autologous plasmablasts engineered to express α-L-iduronidase (IDUA) using the Sleeping Beauty transposon system.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Mucopolysaccharidosis type IH (MPS IH, Hurler syndrome)
* Underwent a previous hematopoietic stem cell transplant >1 year prior to study enrollment
* Age ≥3 years and ≤8 years at time of study registration
* ≥ 10 kilograms body weight
* Creatinine <1.5 normal for gender and age.
* Ejection fraction ≥ 40% by echocardiogram
* Must commit to traveling to the University of Minnesota for the necessary followup evaluations
* Must agree to stay in the Twin Cities area (<45-minute drive from the Masonic Children's Hospital) for a minimum of 5 days after each cell infusion
* Voluntary written parental consent prior to the performance of any study related procedures

Exclusion Criteria:

* Prior enzyme replacement therapy within 4 months prior to enrolling on study
* History of B cell related cancer, EBV lymphoproliferative disease or autoimmune disorders
* Evidence of active graft vs. host disease
* Requirement for systemic immune suppression
* Requirement for continuous supplemental oxygen
* Any medical condition likely to interfere with assessment of safety or efficacy of the study treatment.
* In the investigator's judgement, the subject is unlikely to complete all protocol required study visits or procedures, including follow up visits, or comply with the study requirements for participation.

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2022-12 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 1 Year
  Maximum tolerated dose (MTD) of autologous plasmablasts engineered to express large amounts of α-L-iduronidase (IDUA) using a Sleeping Beauty transposon approach
Growth Velocity (cm/year) | 1 Year
  Growth velocity in centimeters/year over a one-year period through determinations of sitting and standing height at baseline and post infusion
Safety and Tolerability after Infusion: Incidence of Adverse Events | 1 Year
  Incidence of Adverse Events

SECONDARY OUTCOMES:
Z-score Growth Rate | 1 Year
  Estimate the 1-year Z-score growth rate standardized for age and gender
Donor Engraftment | Baseline, 6 months and 1 Year
  Estimate percent myeloid donor chimerism (CD33/66b) at baseline and at 6 and 12 months.
Levels of circulating antibodies (IgG, IgM, IgA and IgE) | 1 Year
  Determine levels of circulating antibodies (IgG, IgM, IgA and IgE) at baseline and at scheduled time points post infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Orchard, MD, Principal Investigator — University of Minnesota, Department of Pediatrics